CLINICAL TRIAL: NCT00830024
Title: A Relative Bioavailability Study of 3 mg Alprazolam Extended Release Tablets Under Non-fasting Conditions
Brief Title: Alprazolam Extended-Release 3mg Tablets Bioequivalence Study Under Non-fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R05-0167
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alprazolam (test) (Experimental): Alprazolam 3 mg ER Tablet (test) dosed in first period followed by Xanax XR® 3 mg Tablet (reference) dosed in second period
  Interventions: Drug: Alprazolam Extended-Release 3 mg Tablets
- Xanax XR® (Active Comparator): Xanax XR® 3 mg Tablet (test) dosed in first period followed by Alprazolam 3 mg ER Tablet (test) dosed in second period
  Interventions: Drug: Alprazolam Extended-Release 3 mg Tablets

INTERVENTIONS:
Drug: Alprazolam Extended-Release 3 mg Tablets — 1 x 3 mg, single dose non-fasting
  Arms: Alprazolam (test)
Drug: Alprazolam Extended-Release 3 mg Tablets — 1 x 3 mg, single dose non-fasting
  Other Names: XANAX XR®
  Arms: Xanax XR®

SUMMARY:
This study will compare the relative bioavailability (rate and extent of absorption) of 3 mg Alprazolam Extended Release Tablets manufactured and distributed by TEVA Pharmaceuticals USA with that of 3 mg XANAX XR® Tablets by Pharmacia & Upjohn Company following a single oral dose (1 x 3 mg extended release tablet) in healthy adult subjects administered under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All subjects selected for this study will be healthy non-smoking men and women 18 years of age or older at the time of dosing. The subject's body mass index (BMI) should be less than or equal to 30.
* Screening procedures: Each subject will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.
* Screening will include general observations, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature. The physical examination will include, but may not be limited to an evaluation of the cardiovascular, gastrointestinal, respiratory, and central nervous systems.

The screening clinical laboratory procedures will include:

* Hematology: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count;
* Clinical Chemistry: serum creatinine, BUN, glucose, AST(GOT), ALT(GPT), albumin, total bilirubin, total protein, and alkaline phosphatase;
* HIV antibody, hepatitis B surface antigen, hepatitis C antibody screens;
* Urinalysis: by dipstick; full microscopic examination if dipstick positive; and
* Urine Drug Screen: ethyl alcohol, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates, and phencyclidine.
* Serum Pregnancy Screen (female subjects only)
* FSH (to verify postmenopausal status; female subjects only)

If female and:

* is postmenopausal for at least 1 year and has a serum FSH level ≥ 20mIU/mL; or
* is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Subjects with a recent history of dug or alcohol addiction or abuse.
* Subjects with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators).
* Subjects whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Subjects demonstrating a reactive screen for hepatitis B surface antigen, hepatitis C antibody or HIV antibody.
* Subjects demonstrating positive drug abuse screen when screened for this study.
* Female subjects demonstrating a positive pregnancy screen.
* Female subjects who are currently breast-feeding.
* Subjects with a history of allergic response(s) to alprazolam or related drugs.
* Subjects with a history of clinically significant allergies including drug allergies.
* Subjects with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Subjects who currently use or report using tobacco products within 90 days of Period I dose administration.
* Subjects who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
* Subjects who report donating greater than 150 mL of blood within 30 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study.
* Subjects who report receiving any investigational drug within 28 days prior to Period I dosing.
* Subjects who report taking any systemic prescription medication in the 14 days prior to Period I dosing.
* Subjects who report an intolerance of direct venipuncture.
* Subjects who report consuming an abnormal diet during the 28 days prior to Period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Carlson, Pharm. D., Principal Investigator — PRACS Institute, Ltd.
Locations (2):
- United States (2):
  - PRACS Institute, Ltd., East Grand Forks, Minnesota
  - PRACS Institute, Ltd., Fargo, North Dakota

RESULTS

PARTICIPANT FLOW:
Groups:
- Test First: Alprazolam Extended Release Tablet 3 mg test product dosed in first period followed by Xanax XR® Tablet 3 mg reference product dosed in second period
- Reference First: Xanax XR® Tablet 3 mg reference product dosed in first period followed by Alprazolam Extended Release Tablet 3 mg test product dosed in second period
Period: First Intervention
Arm/Group | Test First | Reference First
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Washout: 7 Days
Arm/Group | Test First | Reference First
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Test First | Reference First
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test First | Reference First | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 17 | 17 | 34
  Black | 0 | 1 | 1
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Alprazolam: Alprazolam Extended Release Tablet 3 mg test product dosed in either period
- Xanax XR®: Xanax XR® Tablet 3 mg reference product dosed in either period
Arm/Group | Alprazolam | Xanax XR®
Number analyzed (Participants) | 35 | 35
ng/mL | 28.79 (6.35) | 28.95 (5.38)
Statistical Analysis 1: Comparison: Alprazolam vs Xanax XR®; Test type: Non-Inferiority or Equivalence — An analysis of variance (ANOVA) was performed on each of the pharmacokinetic parameters using SAS® software; Geometric Test/Ref Ratio x 100 = 98.75, 90% CI [93.35 to 104.47] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Alprazolam | Xanax XR®
Number analyzed (Participants) | 35 | 35
ng*h/mL | 650.91 (249.36) | 683.25 (289.69)
Statistical Analysis 1: Comparison: Alprazolam vs Xanax XR®; Test type: Non-Inferiority or Equivalence — An analysis of variance (ANOVA) was performed on each of the pharmacokinetic parameters using SAS® software; Geometric Test/Ref Ratio x 100 = 95.94, 90% CI [91.76 to 100.3] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 72 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Alprazolam | Xanax XR®
Number analyzed (Participants) | 35 | 35
ng*h/mL | 600.24 (199.80) | 626.54 (216.46)
Statistical Analysis 1: Comparison: Alprazolam vs Xanax XR®; Test type: Non-Inferiority or Equivalence — An analysis of variance (ANOVA) was performed on each of the pharmacokinetic parameters using SAS® software; Geometric Test/Ref Ratio x 100 = 95.89, 90% CI [91.67 to 100.31] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.